CLINICAL TRIAL: NCT05840601
Title: Evaluation of Dexterous Terminal Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant concluded.
Sponsor: Liberating Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Device Feasibility
Other Study IDs: 271065
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Amputation; Amputation, Traumatic; Amputation; Traumatic, Hand; Limb; Absence, Congenital, Upper; Prosthesis User; Upper Limb Amputation Below Elbow (Injury); Upper Limb Amputation At the Hand
Keywords: amputee; upper limb amputee; upper limb prosthesis user; prosthesis; upper limb absence; dexterous fingertip; index finger prosthesis
MeSH Terms: conditions — Amputation, Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: In the lab, a functional test will be used to evaluate the feasibility of the device design as compared with a baseline condition. A subset of these subjects will test the investigational device at home for up to 2 weeks to provide feedback on the investigational device when used in everyday tasks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pointdexter (Experimental): The investigational device being tested is Pointdexter, a novel prosthetic finger with a built-in split gripper. The device is an index finger which can drop in place of existing fingers on a prosthetic hand. The investigational device is controlled with the same signals used to control the hand. Participants will use a commercially available prosthetic hand compatible with the Pointdexter device for this study.
  Interventions: Device: Pointdexter
- Comparator (Active Comparator): The comparator device is the same commercially available hand that is being used for the Pointdexter arm, except that it will be unmodified (i.e., it will have its usual index finger attached instead of the Pointdexter finger).
  Interventions: Device: Comparator

INTERVENTIONS:
Device: Pointdexter — Commercially available prosthetic hand modified with the investigational Pointdexter finger in place of the usual index finger.
  Other Names: Dexterous Terminal Device
  Arms: Pointdexter
Device: Comparator — Unmodified commercially available prosthetic hand.
  Arms: Comparator

SUMMARY:
Liberating Technologies, Inc. (LTI) has developed Pointdexter, a dexterous prosthetic fingertip that is integrated into a commercial prosthetic hand and allows for an additional fine grasp. The Pointdexter device interfaces with upper limb prostheses by swapping the usual prosthetic pointer finger with the Pointdexter device. The dexterous prosthetic fingertip utilizes the same control strategy used to operate the prosthetic hand. This solution aims to combine the advantages of the common terminal devices into one product by combining the practicality and dexterity of a split-hook or gripper with the aesthetics of multi-articulating hands.

DETAILED DESCRIPTION:
Liberating Technologies, Inc. (LTI) has developed Pointdexter, a dexterous prosthetic fingertip that is integrated into a commercial prosthetic hand and allows for an additional fine grasp. The Pointdexter device interfaces with upper limb prostheses by swapping the usual prosthetic pointer finger with the Pointdexter device. The dexterous prosthetic fingertip utilizes the same control strategy used to operate the prosthetic hand. This solution aims to combine the advantages of the common terminal devices into one product by combining the practicality and dexterity of a split-hook or gripper with the aesthetics of multi-articulating hands.

The rationale for this study is to pilot test the dexterous prosthetic fingertip and gather user feedback. We will conduct in-lab testing to compare the functional outcomes of a commercial prosthetic hand with and without integration of the investigational dexterous fingertip prosthesis. A subset of subjects will take home the device for up to 2 weeks to test out the functionality in their daily lives and provide further feedback. This will be an exploratory pilot study with the intention of gaining a better understanding of device operation throughout activities of daily living (ADLs). User feedback will be collected to inform further development and design.

The study will focus on design feasibility testing and will compare performance of hand functional outcome tests on a commercially available prosthetic hand with and without the investigational Pointdexter modification. Our primary hypothesis is that subjects using the investigational device will show better performance on objective functional outcomes measures than those using a standard prosthetic hand, particularly in the manipulation of small objects.

The investigators will explore multiple outcomes measures as options, but our primary endpoint will be performance on the Small Common Objects subtask of the Jebsen-Taylor Hand Function Test, which assesses a broad range of unimanual hand functions required for ADLs. The primary quantitative measure of the Jebsen-Taylor task will be completion time of each subtask. Myoelectric prosthetic hand users will be recruited for the study and consented with an approved protocol. Able-bodied participants will be recruited for this study as long as they are willing to complete the approved protocol with an upper-limb prosthesis bypass.

There will be one site visit at LTI in Holliston, MA for in-lab functional outcome measure testing. The subject may be asked to return to the lab if testing and/or data collection is incomplete. At the start of the study session, subjects will prepare for testing in their first configuration (investigational or comparator). If investigational, subjects will doff their prosthesis and investigators will replace the usual index finger of the commercially available prosthetic hand being tested with the investigational device. If comparator, subjects will don the unmodified commercially available prosthetic hand. Subjects will be trained on how to operate the investigational device and be allowed a minimum of 30 minutes to practice using it until they are comfortable with proceeding. The subjects will be guided to conduct functional outcome tests that involve picking up and manipulating everyday objects (beans, coins, pegs, spoon, cloth, etc.), such as the tasks outlined in the Jebsen-Taylor and Peg Board functional tests. Each sub-task in the functional test will be scored by occupational therapist standards. After a round of functional testing is done, subjects will fill out a subjective questionnaire. Subjects will then doff the prosthesis and don the next device configuration. Subjects will repeat the functional tests and questionnaire with each device configuration. The study session should span about 4 hours.

A subset of subjects will use the investigational device in their daily lives in place of their usual prosthesis for up to 2 weeks and provide feedback of their experiences with the dexterous prosthetic fingertip. To improve subject convenience and expand our pool of subjects, the take-home study is able to be done fully remote by providing the option to consent through secure voice/video calling and shipping the investigational device to/from the subject.

Upper limb myoelectric prosthesis users and able-bodied individuals will be invited to participate in the study. Research participants will schedule a time to conduct the testing and be informed of study details. Participants will be given as much time as needed to review and question the informed consent form before signing.

Two different technologies will be assessed:

* Investigational Device: Commercially available prosthetic hand with dexterous fingertip modification
* Comparator Baseline: Unmodified commercially available prosthetic hand

Upper limb prosthesis users as well as able-bodied individuals will be recruited for this study through the LTI clinician network and subject database. Prosthetists may be contacted to recruit research subjects and, if interested, will be given flyers to hand out to their patients. If subjects are interested in participating, they can call the number on the flyer to speak with investigators. In addition, previous research participants who have given their permission to be contacted for future studies may be contacted directly to assess their interest in participating in this study.

Based on subject population and availability, a convenience sample of 10 subjects will be recruited for this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Have an upper limb absence
* Uses myoelectric control for their prosthesis
* If they have a major upper limb absence, must use a quick-disconnect wrist
* If able-bodied, must be willing to use an upper-limb prosthesis bypass for testing
* Willing and able to complete activities outlined in the study and provide requested feedback.
* Adults must be able to provide their own consent.

Exclusion Criteria:

* The risks to pregnant people and fetuses are unknown and therefore those who are pregnant should not participate in the study and will be screened by self-disclosure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Jebsen-Taylor Small Common Objects Functional Test | 4 hours
  During the in-lab portion of the study, subjects will be asked to complete the 'small common objects' subtask of the Jebsen-Taylor Hand Function Test, which assesses a broad range of unimanual hand functions required for ADLs. The primary quantitative measure of the Jebsen-Taylor task will be completion time of each subtask. This test will be used to evaluate the feasibility of the device design as compared with the unmodified prosthetic hand.

SECONDARY OUTCOMES:
User Feedback | 4 hours
  Investigators will collect feedback about the device design and how the user would compare manipulating common objects with the investigational device vs. a commercially available prosthetic hand.

IPD SHARING:
Plan to Share IPD: No
Study withdrawn - no participants recruited and no data collected.

REFERENCES:
- See also: Presentation - Initial Clinical Evaluation of Pointdexter - A Dexterous Prosthetic Fingertip — https://figshare.com/articles/poster/Initial_Clinical_Evaluation_of_Pointdexter_-_A_Dexterous_Prosthetic_Fingertip/12792176?file=24384623